CLINICAL TRIAL: NCT06113276
Title: Quantitative Computed Tomography for Mortality Risk Stratification in ARDS
Acronym: CT4ARDS-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0664; 194_v3 (Registry Identifier: CNIL)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; computed tomography; alveolar recruitment; PEEP; tidal hyperinflation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- tidal hyperinflation: As the study aim to identify whether tidal hyperinflation is an independent predictor for ARDS mortality, and as this variable will be entered as a quantitative predictor in the multivariate model, the study encompass a single group of patient (i.e. all included patients)
  Interventions: Radiation: Low dose computed tomography to evaluate biomechanical parameters in the lung

INTERVENTIONS:
Radiation: Low dose computed tomography to evaluate biomechanical parameters in the lung — In the participating to the study, response to PEEP increase and tidal inflation are evaluated with a software computing biomechanical parameters (tidal hyperinflation and lung recruitability). Tidal hyperinflation and recruitment are computed on CT images acquired within 72 hours after ARDS onset or with 72h after ECMO onset.

SUMMARY:
Acute respiratory distress syndrome remains a deadly disease with hospital mortality remaining between 40 to 50%. ARDS mortality risk factors have been identified from patient history, common clinical and biological variables in the lung SAFE study. Part of ARDS mortality is attributable to ventilator-induced lung injury (VILI), in relation with inappropriate settings on the ventilator. Tidal hyperinflation and recruitment/derecruitment during lung inflation are 2 identified mechanisms leading to VILI, that may be identified on computed tomography while poorly identified with variables collected at the bedside.

The aim of this study is to identify whether tidal hyperinflation identified on computed tomography is a risk factor for ARDS mortality, independently from know bio-clinical risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 15 or older with ARDS according to the Berlin definition
* invasive mechanical ventilation with PaO2/FiO2 ≤ 300 mm Hg
* with computed tomography acquired at both end-expiration and end-inspiration, or at both PEEP 5 and 15 cm H2O at end-expiration
* PEEP setting according to a PEEP/FiO2 table, with secondary adjustment according to hemodynamic tolerance
* Tidal volume 6 ml/kg of predicted body weight or less

Exclusion Criteria:

* Use of contrast agent during computed tomography acquisition
* ARDS criteria onset since more than 72 hours or ECMO onset since more than 72 hours
* Proven COPD
* Pneumothorax or bronchopleural fistula
* Patient with spontaneous breathing preventing realization of end-expiratory and end-inspiratory pauses
* Previous inclusion in current study
* Patient under a legal protective measure

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be screened from the population of patient hospitalized for ARDS in the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Odd ratio of tidal hyperinflation assessed on CT at day-0 as an independent predictor of 90-day mortality | Day-0 (time of realization of CT scan)
  Tidal hyperinflation is computed as the volume difference of hyperinflated lung (i.e., with CT attenuation between -1000 and -900 Hounsfield units) between and-expiration and end-inspiration at the PEEP level chosen by clinician

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de Médecine Intensive Réanimation Hôpital Michallon - CHU Grenoble Alpes, La Tronche
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse - Service de Médecine Intensive Réanimation, Lyon
  - Service de Réanimation Polyvalente Centre Hospitalier Lyon Sud Hospices Civils de Lyon, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes, Rennes

REFERENCES:
- [Derived] Shekarnabi M, Guillien A, Terzi N, Sigaud F, Bitker L, Roux E, Ahaouari T, Serrano EED, Boussel L, Ferretti G, Yonis H, Mezidi M, Noirot I, Chauvelot L, Dhelft F, Gaillet M, Siroux V, Orkisz M, Richard JC, Bayat S. Prognostic value of functional CT imaging in COVID-ARDS: a two-centre prospective observational study. Respir Res. 2025 May 9;26(1):177. doi: 10.1186/s12931-025-03232-7. PMID 40346553